CLINICAL TRIAL: NCT06413771
Title: Comparison of Two Ovarian Stimulation Strategies in Intrauterine Insemination Cycles of Couples With Unexplained Infertility; Only Gonadotropin Vs. Letrozole Combined Gonadotropin Stimulation. A Randomized Controlled Trial.
Brief Title: Only Gonadotropin Vs. Letrozole Combined Gonadotropin Stimulation in IUI Cycles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, GÜRKAN UNCU,PROF. MD, Prof., Uludag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-4/39
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Infertility Unexplained
Keywords: unexplained infertility; letrozole; gonadotropin; intrauterine insemination
MeSH Terms: interventions — Letrozole; Gonadotropins

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Patients were divided into two study arms based on the initial digits of their national IDs by ART nurses. Importantly, the IVF clinicians remained blinded to the patients' grouping throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Only Gonadotropin (Active Comparator): The Conventional Only Gonadotropin (COG) group received recombinant FSH based on body mass index (BMI)
  Interventions: Drug: Gonadotropin
- Combined Letrozole-Gonadotropin group (Active Comparator): The combined Letrozole-Gonadotropin (CLG) group received letrozole followed by gonadotropin with dose adjustments based on BMI.
  Interventions: Drug: Letrozole 2.5mg

INTERVENTIONS:
Drug: Letrozole 2.5mg — Letrozole pretreatment during ovarian stimulation with gonadotropins, in intrauterine insemination cycles.
  Arms: Combined Letrozole-Gonadotropin group
Drug: Gonadotropin — Ovarian stimulation with gonadotropins, in intrauterine insemination cycles.
  Arms: Conventional Only Gonadotropin

SUMMARY:
The present randomized controlled study aims to investigate the effectiveness of a combined regimen of letrozole and gonadotropin with dose adjustments based on body mass index (BMI) compared to a conventional only gonadotropin regimen in intrauterine insemination (IUI) cycles for couples experiencing unexplained infertility. The study was conducted at a tertiary university hospital's Assisted Reproductive Technologies (ART) center from January 2023 to January 2024. Couples with unexplained infertility were enrolled based on comprehensive assessments, and randomization was performed based on national ID (odd or even). The Conventional Only Gonadotropin (COG) group received recombinant FSH based on body mass index (BMI), while the Combined Letrozole-Gonadotropin (CLG) group received letrozole followed by gonadotropin with dose adjustments based on BMI. Ovulation induction and IUI were performed according to standard protocols. Clinical outcomes, gonadotropin consumption, and pregnancy rates were compared between groups. Among 317 IUI cycles, 131 couples with unexplained infertility were randomized (CLG: 61, COG: 70). Demographic parameters were similar between groups. The CLG group had lower daily gonadotropin doses (67 ± 18 IU/D vs. 76 ± 11 IU/d, p=0.01) and total gonadotropin consumption (750 IU vs. 825 IU, p=0.01) with comparable ovulation and clinical pregnancy rates. The COG group exhibited higher multiple pregnancy rates, although not statistically significant (CLG vs. COG; 1/61 vs. 3/70, p=0.4). The study suggests that the combined letrozole and gonadotropin regimen with BMI-based dose adjustments in IUI cycles for unexplained infertility is associated with reduced gonadotropin consumption and potentially lower multiple pregnancy rates.

ELIGIBILITY:
Inclusion Criteria:

* Couples with unexplained infertility
* Aged between 18-35

Exclusion Criteria:

* Male factor infertility
* Diminished ovarian reserve
* Patient refusion to participate

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 131 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Clinical Pregnancy Rate | 6 weeks
  Presence of gestational sac by transvaginal ultrasound

SECONDARY OUTCOMES:
Multiple Pregnancy Rate | 6 weeks
  Presence of multipl gestational sacs by transvaginal ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Gurkan Uncu, Prof., Study Chair — Uludag University
Locations (1):
- Uludag University Faculty of Medicine, Bursa, Gorukle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
All data generated or analyzed during this study are included in this published article and are available from the corresponding author on reasonable request.